CLINICAL TRIAL: NCT05845047
Title: PICTURE IT: Producing Increasingly Complex Themes Using Right-hemisphere Engagement (PICTURE) Implemented With Telemedicine
Brief Title: Producing Increasingly Complex Themes Using Right-hemisphere Engagement (PICTURE) Implemented With Telemedicine
Acronym: PICTURE IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00387816
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study is to be conducted in a blinded assessor manner. The participants and the clinician performing the behavioral assessments will know the treatment assignment, as there is no way to mask the participants from this information. The PI will have access to the unblinded list of randomization codes and treatment assignments. Technicians who were not involved in any of the treatment sessions will review videos of all of the assessments and will score the participants without knowledge of treatment order assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICTURE IT Intervention-CoDeLT Intervention (Experimental): Participants will receive PICTURE IT Intervention for 15 sessions followed by Computer Delivered Lexical Treatment (CoDeLT)Intervention for 15 sessions
  Interventions: Behavioral: PICTURE-IT; Behavioral: CoDeLT
- CoDeLT Intervention-PICTURE IT Intervention (Active Comparator): Participants will receive Computer Delivered Lexical Treatment (CoDeLT) Intervention for 15 sessions followed by PICTURE IT Intervention for 15 sessions
  Interventions: Behavioral: PICTURE-IT; Behavioral: CoDeLT

INTERVENTIONS:
Behavioral: PICTURE-IT — The speech-language pathologist (SLP) will provide one of the following stimuli hierarchically:
  1. Single words depicted in the picture, then with written and spoken labels
  2. 2-word phrases depicted in the picture and then with written and spoken word
  3. Subject-Verb-Object sentence depicted in the picture and then with written and spoken sentences
  4. Two-sentence event, depicted with photos and subsequently with two written and spoken sentences
  5. Short story depicted with a video clip and subsequently with printed and spoken narrative.
  Sessions will be completed online with a speech-language pathologist using video conferencing software, using a laptop and a hot spot the investigators will provide if needed. Participants in both groups will receive the same 15 45-minute sessions of a PICTURE-IT.
  Other Names: Producing Increasingly Complex Themes Using Right-hemisphere Engagement Implemented with Telemedicine
Behavioral: CoDeLT — The speech-language pathologist (SLP) will facilitate the computer-delivered naming treatment, consisting of a picture/seen and heard spoken word verification task.
  A picture will be presented for two seconds on a laptop computer screen and will be immediately followed by an audio-visual display of a speaker's mouth saying a noun, phrase, or sentence. The spoken word, phrase, or sentence either will or will not fit the preceding picture, and the participant must indicate whether the picture and video match or do not match. The computer will provide immediate visual feedback following a response.
  Sessions will be completed online with a speech-language pathologist using video conferencing software, using a laptop and a hot spot the investigators will provide if needed. Participants in both groups will receive the same 15 45-minute sessions of a PICTURE-IT.
  Other Names: Computer Delivered Lexical Treatment

SUMMARY:
The investigators propose a pilot crossover trial of 2 behavioral language treatments, with randomized order of treatments and blinded assessors, to determine if a therapy designed to stimulate right hemisphere functions (Producing Increasingly Complex Themes Using Right-hemisphere Engagement Implemented with Telemedicine - PICTURE IT; described below) is more effective in improving discourse than a published computer delivered lexical treatment (shown previously to improve naming) in subacute post-stroke aphasia.

DETAILED DESCRIPTION:
The investigators will carry out a crossover study with randomized order of treatment conditions and blinded assessors, to compare changes in content and efficiency of discourse (primary outcome measures) from before treatment to immediately after treatment, to compare intervention focused on engaging the right hemisphere (PICTURE IT; see below) to a purely lexical treatment (see details below). Secondary outcome measures will be: (1) changes in discourse from pre-treatment to 2 weeks post-treatment, and (2) changes in naming of objects and actions from immediately before treatment to immediately after treatment, and (3) changes in naming of objects and actions from pre-treatment to 2 months after both treatments. The investigators will also carry out resting state functional near infrared spectroscopy (fNIRS) before and after each treatment to evaluate degree and location (e.g. intrahemispheric right versus left) of changes in connectivity associated with each treatment and with changes in each outcome measure. The investigators will also take saliva samples from participants who agree to this optional part of the study to determine the participants brain-derived neurotrophic factor status.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Premorbid proficiency in English
3. Left hemisphere ischemic or hemorrhagic stroke confirmed by imaging, which occurred either 1-4 months or ≥ 6 months ago
4. Diagnosis of aphasia secondary to stroke as defined using the Western Aphasia Battery-Revised Aphasia Quotient < 93.8.
5. Capable of giving informed consent or indicating another to provide informed consent

Exclusion Criteria:

1. Prior history of neurologic disease affecting the brain (e.g., brain tumor, multiple sclerosis, traumatic brain injury) other than stroke
2. Prior history of severe psychiatric illness, developmental disorders or intellectual disability (e.g., PTSD, schizophrenia, obsessive-compulsive disorder, autism spectrum disorders)
3. Inability to follow the treatment procedure as indicated by appropriate (not necessarily accurate) engagement during 5 probes of each.
4. Uncorrected severe visual loss or hearing loss by self-report and medical records

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2031-08 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Change in discourse content as assessed by z-score for the number of meaning-carrying units used in describing a picture | Baseline, 1 week after treatment
  Change in z-score for the number of meaning-carrying units used in describing a picture. There is no maximum number of meaning-carrying units, but norms are available to assist in the interpretation of this performance.

SECONDARY OUTCOMES:
Change in discourse informational efficiency as assessed by z-score for the number of syllables of meaning-carrying units used in describing a picture | Baseline, 1 week after treatment
  Change in z-score for the number of syllables/number of meaning-carrying units used in describing a picture. There is no maximum number of meaning-carrying units, but norms are available to assist in the interpretation of this performance.
Change in accuracy of naming objects as assessed by the Boston Naming Test | Baseline, 1 week after treatment
  Change in accuracy of naming objects on the 30-item Boston Naming Test. Scores range from 0 to 30 with higher scores meaning better naming ability.
Change in accuracy of naming actions as assessed by the Hopkins Action Naming Assessment form | Baseline, 1 week after treatment
  Change in accuracy of naming actions on the 30-item Hopkins Action Naming Assessment. Scores range from 0 to 30 with higher scores meaning better naming ability.
Change in resting state functional connectivity as assessed by near-infrared spectroscopy | Baseline, 1 week after treatment
  Measure of correlation between activation of brain regions at rest using functional near-infrared spectroscopy. Right hemisphere intrahemispheric, left hemisphere intrahemispheric, and interhemispheric measures will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Argye E Hillis, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert ML, Sparks RW, Helm NA. Melodic intonation therapy for aphasia. Arch Neurol. 1973 Aug;29(2):130-1. doi: 10.1001/archneur.1973.00490260074018. No abstract available. PMID 4717723
- [Background] Baker JM, Rorden C, Fridriksson J. Using transcranial direct-current stimulation to treat stroke patients with aphasia. Stroke. 2010 Jun;41(6):1229-36. doi: 10.1161/STROKEAHA.109.576785. Epub 2010 Apr 15. PMID 20395612
- [Background] Berube S, Nonnemacher J, Demsky C, Glenn S, Saxena S, Wright A, Tippett DC, Hillis AE. Stealing Cookies in the Twenty-First Century: Measures of Spoken Narrative in Healthy Versus Speakers With Aphasia. Am J Speech Lang Pathol. 2019 Mar 11;28(1S):321-329. doi: 10.1044/2018_AJSLP-17-0131. PMID 30242341
- [Background] Breining BL, Faria AV, Caffo B, Meier EL, Sheppard SM, Sebastian R, Tippett DC, Hillis AE. Neural regions underlying object and action naming: Complementary evidence from acute stroke and primary progressive aphasia. Aphasiology. 2022;36(6):732-760. doi: 10.1080/02687038.2021.1907291. Epub 2021 May 11. PMID 35832655
- [Background] Crosson B, Moore AB, Gopinath K, White KD, Wierenga CE, Gaiefsky ME, Fabrizio KS, Peck KK, Soltysik D, Milsted C, Briggs RW, Conway TW, Gonzalez Rothi LJ. Role of the right and left hemispheres in recovery of function during treatment of intention in aphasia. J Cogn Neurosci. 2005 Mar;17(3):392-406. doi: 10.1162/0898929053279487. PMID 15814000
- [Background] Crosson B, Moore AB, McGregor KM, Chang YL, Benjamin M, Gopinath K, Sherod ME, Wierenga CE, Peck KK, Briggs RW, Rothi LJ, White KD. Regional changes in word-production laterality after a naming treatment designed to produce a rightward shift in frontal activity. Brain Lang. 2009 Nov;111(2):73-85. doi: 10.1016/j.bandl.2009.08.001. Epub 2009 Oct 6. PMID 19811814
- [Background] Fridriksson J, Elm J, Stark BC, Basilakos A, Rorden C, Sen S, George MS, Gottfried M, Bonilha L. BDNF genotype and tDCS interaction in aphasia treatment. Brain Stimul. 2018 Nov-Dec;11(6):1276-1281. doi: 10.1016/j.brs.2018.08.009. Epub 2018 Aug 18. PMID 30150003
- [Background] Mack WJ, Freed DM, Williams BW, Henderson VW. Boston Naming Test: shortened versions for use in Alzheimer's disease. J Gerontol. 1992 May;47(3):P154-8. doi: 10.1093/geronj/47.3.p154. PMID 1573197
- [Background] Popescu T, Stahl B, Wiernik BM, Haiduk F, Zemanek M, Helm H, Matzinger T, Beisteiner R, Fitch WT. Melodic Intonation Therapy for aphasia: A multi-level meta-analysis of randomized controlled trials and individual participant data. Ann N Y Acad Sci. 2022 Oct;1516(1):76-84. doi: 10.1111/nyas.14848. Epub 2022 Aug 2. PMID 35918503
- [Background] Saur D, Lange R, Baumgaertner A, Schraknepper V, Willmes K, Rijntjes M, Weiller C. Dynamics of language reorganization after stroke. Brain. 2006 Jun;129(Pt 6):1371-84. doi: 10.1093/brain/awl090. Epub 2006 Apr 25. PMID 16638796